CLINICAL TRIAL: NCT07056881
Title: Monotherapy vs Combination Therapy for Bone Infections Caused by Pseudomonas Aeruginosa
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0108_REANIMATION_OPERA
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Osteomyelitis; Pseudomonas Infections; Pseudomonas Aeruginosa; Bacterial Infections
MeSH Terms: conditions — Osteomyelitis; Pseudomonas Infections; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at how well one antibiotic (monotherapy) works compared to two antibiotics (combination therapy) in treating bone infections caused by Pseudomonas aeruginosa. It includes 300 adult patients who had this type of infection confirmed by lab tests and medical imaging. The goal is to find out if using just one antibiotic is as effective as using two, while also looking at side effects, the need for more surgery, antibiotic resistance, and overall antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Diagnosis of osteitis or osteomyelitis due to Pseudomonas aeruginosa
* Isolation of Pseudomonas aeruginosa from at least one deep, sterile sample (e.g., bone biopsy, joint aspiration)
* Imaging findings consistent with osteomyelitis (MRI, CT scan, or X-ray)

Exclusion Criteria:

* No isolation of Pseudomonas aeruginosa
* No imaging evidence suggestive of osteomyelitis
* Patients under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the electronic health records of adult patients hospitalized within the AP-HP (Assistance Publique-Hôpitaux de Paris) network. The study population includes individuals diagnosed with osteitis or osteomyelitis who have a confirmed microbiological diagnosis of Pseudomonas aeruginosa infection, along with imaging consistent with bone infection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate at the end of antibiotic treatment, defined as resolution of signs and symptoms of infection without need for additional antibiotic therapy or surgical intervention. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France, France